CLINICAL TRIAL: NCT05929079
Title: A Master Protocol to Investigate the Efficacy and Safety of LY3437943 Once Weekly in Participants With Type 2 Diabetes Mellitus Who Have Obesity or Overweight: A Randomized Double-Blind, Placebo-Controlled Trial
Brief Title: A Study of Retatrutide (LY3437943) in Participants With Type 2 Diabetes Mellitus Who Have Obesity or Overweight
Acronym: TRIUMPH-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18558; J1I-MC-GZBK (Other: Master Protocol Eli Lilly and Company); J1I-MC-GSA2 (Other: ISA Eli Lilly and Company); 2023-503658-11-00 (Other: EU Trial Number)
Record Dates: First submitted 2023-06-26; First posted 2023-07-03 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes; Obesity; Overweight; Obstructive Sleep Apnea
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Overweight; Sleep Apnea, Obstructive | interventions — retatrutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Retatrutide Dose 1 (Experimental): Participants will receive retatrutide subcutaneously (SC).
  Interventions: Drug: Retatrutide
- Retatrutide Dose 2 (Experimental): Participants will receive retatrutide SC.
  Interventions: Drug: Retatrutide
- Retatrutide Dose 3 (Experimental): Participants will receive retatrutide SC.
  Interventions: Drug: Retatrutide
- Placebo (Placebo Comparator): Participants will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Retatrutide — Administered SC
  Other Names: LY3437943
  Arms: Retatrutide Dose 1; Retatrutide Dose 2; Retatrutide Dose 3
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to is to evaluate the efficacy and safety of retatrutide in participants with type 2 diabetes in participants who have obesity or overweight (J1I-MC-GZBK master protocol) including a subset of participants who have obstructive sleep apnea (OSA) (J1I-MC-GSA2). The study will last about 89 weeks and will include up to 24 visits.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) greater than or equal to 27.0 kilogram/square meter (kg/m ²)
* Have Type 2 Diabetes (T2D)
* Are on stable treatment for T2D for at least 90 days
* Have a history of at least one unsuccessful dietary effort to lose body weight.

GSA2 Inclusion Criteria

* Previously diagnosed with OSA
* Have AHI ≥15 on polysomnography at screening (definition of moderate-to-severe OSA)
* For participants not on positive airway pressure (PAP) therapy: unable or unwilling to use PAP therapy and have not used PAP for at least 4 weeks prior to screening.
* If on PAP therapy, have been on PAP therapy for at least 3 consecutive months prior to screening, and willing to temporarily stop using PAP therapy for approximately 7 days prior to each of the sleep study (PSG) visits.

Exclusion Criteria:

* Have a self-reported or documented change in body weight >5 kg (11 pounds) within 90 days.
* Have taken weight loss drugs, including over-the-counter medications, within 90 days prior to screening.
* Have a prior or planned surgical treatment for obesity.
* Have Type 1 diabetes
* Have a family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN-2)
* Have had pancreatitis

GSA2 Exclusion Criteria

* Use stimulants (for example, modafinil, armodafinil, solriamfetol, pitolisant, amphetamine) less than 3 months prior to screening.
* Use hypnotics, mirtazapine, opioids, trazodone, and zonisamide less than 3 months prior to screening.
* Use a dental appliance or other device to treat OSA other than PAP therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline, Week 80
Change from Baseline in Apnea-Hypopnea Index (AHI) for GSA2 Subset | Baseline, Week 80

SECONDARY OUTCOMES:
Change from Baseline in Body Mass Index (BMI) | Baseline, Week 80
Change from Baseline in Waist Circumference | Baseline, Week 80
Change from Baseline in Systolic Blood Pressure (SBP) | Baseline, Week 80
Change from Baseline in Diastolic Blood Pressure (DBP) | Baseline, Week 80
Percent Change from Baseline in Total Cholesterol | Baseline, Week 80
Percent Change from Baseline in Triglycerides | Baseline, Week 80
Change from Baseline in Hemoglobin (A1c) HbA1c % | Baseline, Week 80
Change from Baseline in Short Form 36 Version 2 (SF-36v2) Acute Form Physical Functioning Domain Score | Baseline, Week 80
Change from Baseline in Fasting Glucose | Baseline, Week 80
Pharmacokinetics (PK): Steady State Area Under the Concentration Time Curve (AUC) | Baseline through Week 80
  AUC is presented as a single average measure of AUC across the study duration.
Percent Change from Baseline in Apnea-Hypopnea Index (AHI) for GSA2 Subset | Baseline, Week 80
A Hierarchical Combination of Functional Outcomes of Sleep Questionnaire (FOSQ) 10 score, FOSQ Vigilance Domain Score, and FOSQ Activity Level Domain Score for GSA2 Subset | Baseline to Week 80
  A hierarchical combination of change from baseline in the FOSQ 10 score, FOSQ Vigilance Domain Score, and FOSQ Activity Level Domain Score will be assessed by the win ratio. The reported unit will be the total "wins" for each treatment group from performing a hierarchical comparison of the component.
Percentage of Participants with ≥50% AHI Reduction from Baseline for GSA2 Subset | Baseline to Week 80
Percentage of Participants with AHI <5 or with AHI 5-14 with Epworth Sleepiness Scale (ESS) ≤10 for GSA2 Subset | Week 80

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (98):
- United States (40):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Cullman Clinical Trials, Cullman, Alabama
  - Preferred Research Partners, Little Rock, Arkansas
  - Core Healthcare Group, Cerritos, California
  - Velocity Clinical Research, Westlake, Los Angeles, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Teradan Clinical Trials, LLC, Brandon, Florida
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - Therafirst Medical Center, Fort Lauderdale, Florida
  - Clinical Site Partners LLC, dba Flourish Research, Miami, Florida
  - Quantum Clinical Trials, Miami Beach, Florida
  - Renstar Medical Research, Ocala, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Clinical Site Partners, LLC dba Flourish Research, Winter Park, Florida
  - NeuroTrials Research Inc, Atlanta, Georgia
  - Centricity Research Rincon Pulmonology, Rincon, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Brengle Family Medicine, Indianapolis, Indiana
  - MedVadis Research Corporation, Waltham, Massachusetts
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Mid Hudson Medical Research, New Windsor, New York
  - Monroe Biomedical Research, Monroe, North Carolina
  - Carteret Medical Group, Morehead City, North Carolina
  - Lillestol Research, Fargo, North Dakota
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Intrepid Research, Cincinnati, Ohio
  - Preferred Primary Care Physicians, Preferred Clinical Research (Ofc 18), Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - Trial Management Associates, Myrtle Beach, South Carolina
  - Tribe Clinical Research - Spartanburg, Spartanburg, South Carolina
  - FutureSearch Trials of Neurology, Austin, Texas
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - Advanced Research Institute, Ogden, Utah
  - Northwest Clinical Research Center, Bellevue, Washington
- Argentina (4):
  - Consultorio de Investigación Clínica EMO SRL, Buenos Aires, Buenos Aires F.D.
  - Centro Médico Viamonte, Buenos Aires, Buenos Aires F.D.
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires, Buenos Aires F.D.
  - Centro de Salud e Investigaciones Médicas, Santa Rosa, La Pampa Province
- Australia (12):
  - Emeritus Research, Botany, New South Wales
  - Woolcock Institute of Medical Research, Macquarie Park, New South Wales
  - The AIM Centre / Hunter Diabetes Centre, Merewether, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Core Research Group, Brisbane, Queensland
  - Nightingale Research, Adelaide, South Australia
  - Flinders University, Bedford Park, South Australia
  - Southern Adelaide Diabetes & Endocrine Services, Oaklands Park, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Emeritus Research, Camberwell, Victoria
  - Austin Health - Repatriation Hospital, Heidelberg West, Victoria
  - Advara HeartCare Joondalup, Joondalup, Western Australia
- Brazil (3):
  - BR Trials - Ensaios Clinicos e Consultoria, São Paulo, São Paulo
  - CPQuali Pesquisa Clínica, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
- India (14):
  - All India Institute of Medical Sciences, Raipur, Chhattisgarh
  - V.S. General Hospital, Ahmedabad, Gujarat
  - Avron Hospitals, Ahmedabad, Gujarat
  - Zydus Hospitals & Healthcare Research Pvt.Ltd., Ahmedabad, Gujarat
  - Life Care Hospital and Research Centre, Bangalore, Karnataka
  - Sushruta Multispeciality Hospital & Research Centre, Hubli, Karnataka
  - Mysore Medical College, Mysore, Karnataka
  - CARE CHL-Hospitals, Indore, Madhya Pradesh
  - Sawai Man Singh Medical College Hospital (SMS Hospital), Jaipur, Rajasthan
  - Madras Diabetes Research Foundation, Chennai, Tamil Nadu
  - Christian Medical College Vellore, Vellore, Tamil Nadu
  - Care Hospitals Hyderabad- Banjara Hills, Hyderabad, Telangana
  - Diabetes Research Center, Hyderabad, Telangana
  - Institute of Post Graduate Medical Education and Research and Seth Sukhlal Karnani Memorial Hospital, Kolkata, West Bengal
- Mexico (12):
  - Centro de Investigacion en Artritis y Osteoporosis SC, Mexicali, Estado de Baja California
  - Diseno y Planeacion en Investigacion Medica, Guadalajara, Jalisco
  - Private Practice - Dr. Arechavaleta Granell Maria del Rosario, Guadalajara, Jalisco
  - Unidad de Investigación Clínica y Atención Médica HEPA, Guadalajara, Jalisco
  - RM Pharma Specialists, Mexico City, Mexico City
  - Clinica Omega, Mexico City, Mexico City
  - Centro Especializado En Diabetes, Obesidad Y Prevencion De Enfermedades Cardiovasculares, Mexico City, Mexico City
  - Cardiolink Clin Trials, Monterrey, Nuevo León
  - Unidad biomedica avanzada monterrey, Monterrey, Nuevo León
  - Investigacion En Salud Y Metabolismo S.C / Nutricion Clinica / Unidad de Base de Datos, Chihuahua City
  - FAICIC S. de R.L. de C.V., Veracruz
  - Arké SMO S.A de C.V, Veracruz
- Romania (6):
  - Diabdana, Oradea, Bihor County
  - Geea Medical Easy Diet, Bucharest, București
  - Centrul Medical NutriLife, Bucharest, București
  - Gama Diamed, Mangalia, Constanța County
  - Centrul Medical Mediab, Târgu Mureş, Mureș County
  - CMI Dr.Pletea Noemi SRL, Bacau
- Spain (7):
  - Centro Periférico de Especialidades Bola Azul, Almería, Almería
  - H.R.U Málaga - Hospital Civil, Málaga, Andalusia
  - Hospital Universitario Virgen de la Victoria, Málaga, Andalusia
  - Complejo Asistencial Universitario de León - Hospital de León, León, Castille and León
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - Vithas Hospital Sevilla, Seville, Sevilla
  - Hospital Universitario Virgen Del Rocio, Seville

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: a are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Retatrutide (LY3437943) in Participants With Type 2 Diabetes Mellitus Who Have Obesity or Overweight (TRIUMPH-2) — https://trials.lilly.com/en-US/trial/408215